CLINICAL TRIAL: NCT06533501
Title: Leucine Requirements During Different Phases of the Menstrual Cycle in Eumenorrheic Women
Brief Title: Leucine Requirements During the Menstrual Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H23-03387
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Menstrual Cycle

STUDY DESIGN:
Intervention Model Description: Single-day interventions; Repeated Measures Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Leucine Intake (Experimental): Randomly assigned one of 7 test leucine intakes that range from deficient to excess (10mg/kg/d to 85mg/kg/d). Participants may complete up to 7 study days in each menstrual phase, at different randomly assigned intakes.
  Interventions: Other: Dietary Leucine Intakes

INTERVENTIONS:
Other: Dietary Leucine Intakes — Participants consume 8 hourly meals that contain the assigned test leucine intake. Each meal will provide one-twelfth of the participants' daily energy requirements as estimated by 1.5 x Resting Energy Expenditure (REE) and adequate protein at 1.0 g.kg.d, to maintain a metabolic steady state. The meals are in the form of a crystalline amino acid protein shake, and protein-free cookies.

SUMMARY:
The existing guidelines for dietary amino acid intake for women are set the same as those established for men. These recommendations might not be appropriate for women, as they do not take into consideration important differences between male and female physiology, like the menstrual cycle. This study aims to determine the leucine requirements during the phases of the menstrual cycle. Leucine is an essential amino acid (cannot be made naturally in the body) and is necessary for protein synthesis, and other important cellular functions. Consuming an adequate amount daily is crucial for maintaining overall health. An innovative, non-invasive technique utilizing pre-determined diets, safe stable isotopes, and a simple breath collection method will be used. Previous work done by Elango Lab investigators has applied this method to investigate other amino acids in pregnant, non-pregnant, and lactating women.

DETAILED DESCRIPTION:
The objective of the study is to determine leucine requirements using the indicator amino acid oxidation method during the follicular phase and the luteal phase of the menstrual cycle in healthy women (between the ages of 20-35 y).In comprehending protein needs and achieving protein targets, it is imperative to establish individual amino acid requirements. This clinical study aims to determine the dietary requirements of leucine for women, helping build a strong foundation for setting dietary guidelines for women. The existing values, derived from guidelines designed for men, overlook the crucial impact of the menstrual cycle on energy and dietary intake. Relying on amino acid requirements derived from studies in men for women significantly heightens the risk of potential harm. It is crucial to identify the distinct amino acid requirements for women and grasp how these needs are affected by various phases of the menstrual cycle. A minimum of 15 healthy women (20-35 y) will be recruited and studied at two menstrual phases over a range of test leucine intakes (10, 20, 30, 40, 55, 70, and 85 mg/kg/day). Women will be invited to participate in up to 7 study days/phase, and randomized to a different intake at each study day. Participants' eligibility will be assessed during a pre-study day. The goal is to study a minimum of 7 women at each intake, for a total of 49 study days in each stage.

ELIGIBILITY:
Inclusion Criteria:

* People with menstrual cycles
* Between the ages of 20 to 35y
* Regular menstrual cycle (21-35 day cycle) for the past 12 months
* Body mass index (BMI) of between 18 and 28 kg/m2
* Free from pre-existing health conditions

Exclusion Criteria:

* People who are currently using hormonal birth control or any contraceptive that would affect sex hormones
* People on hormone therapy
* People with an abnormal menstrual cycle history
* People with non-traditional dietary practices
* Recent weight loss/weight gain
* People with a history of endocrine disorders
* People who are pregnant
* People who are breastfeeding
* People who have given birth in the last 18 months
* People who depend on medication that affects normal metabolism. Any medication that alters normal body metabolism would skew the results and compromise the validity of the data set.
* People with a metabolic, neurological, genetic, or immune disorder likely to affect nutritional requirements or overall body metabolism.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Carbon 13 Oxidation | 8 hours
  Urine and breath samples will be collected to measure the rate of L-[1-13C]phenylalanine oxidation.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada